CLINICAL TRIAL: NCT03108378
Title: A Prospective Multicenter Cohort Study Evaluating the Long Term Retention of Gadolinium in Human Bone and Skin After the Retrospective Administration of MultiHance or ProHance in Comparison With a Control Group Receiving No Exposure to Gadolinium
Brief Title: Evaluation of Gd Retention in Human Bone and Skin After MultiHance or ProHance Administration Compared With Control
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: GMRA-102
Record Dates: First submitted 2017-02-22; First posted 2017-04-11 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Gadolinium Retention
Keywords: Gadolinium; Bone; Skin
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Bone & Skin Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- MultiHance Single Dose: Subjects who received a single dose of MultiHance and no other Gd agent and who are also scheduled for orthopedic surgery
  Interventions: Procedure: Surgery
- MultiHance Multiple Dose: Subjects who received multiple doses of MultiHance and no other Gd agent and who are also scheduled for orthopedic surgery
  Interventions: Procedure: Surgery
- ProHance Single Dose: Subjects who received a single dose of ProHance and no other Gd agent and who are also scheduled for orthopedic surgery
  Interventions: Procedure: Surgery
- ProHance Multiple Dose: Subjects who received multiple doses of ProHance and no other Gd agent and who are also scheduled for orthopedic surgery
  Interventions: Procedure: Surgery
- Control Subgroup: Subjects who have not received any Gd agent and who are also scheduled for orthopedic surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures

SUMMARY:
Subjects must be scheduled to undergo an orthopedic surgical procedure. Subjects in the non-control group must have previously received an MRI with MultiHance or ProHance with at least 1 month between the last administration and the scheduled surgery. Subjects who have never received MultiHance or ProHance or any other gadolinium agent will also be enrolled. Subjects must have a test of their kidney function (SCr) at the time of the last MRI examination or at the time of enrollment if they never received gadolinium.

A sample of bone and skin will be collected from the scheduled surgery and tested for the amount of gadolinium. An additional sample of skin will be collected for testing the presence of nephrogenic systemic fibrosis (NSF).

DETAILED DESCRIPTION:
Each subject enrolled will already be scheduled to undergo a hip, shoulder or knee replacement, limb amputations or other orthopedic surgical procedures and each subject enrolled in the non-control group will have retrospectively undergone one or more administrations of MultiHance or PROHANCE with the last dose administered at least 1 month before their scheduled surgery. In order to classify the subjects' renal status, the serum creatinine (SCr) value and/or estimated glomerular filtration rate (eGFR) at the time of last MRI with MultiHance or ProHance must be available and collected. The control subjects' documented SCr values will be collected prior to enrollment in the study.

The bone and skin tissue sample(s) collected (during the subjects surgery) will be blinded to gadolinium based contrast agent (GBCA) exposure and sent to a central laboratory where they will be tested for gadolinium (Gd) and other analytes including calcium, phosphorous, sodium, iron, zinc, and potassium. The Gd deposition of the resected bone and skin tissue will be analyzed by Inductively Coupled Plasma Mass Spectroscopy (ICP-MS). The bone and skin tissue will also be analyzed for other analytes using ICP-MS. These sample(s) will be stored at the central laboratory.

A separate sample of the skin tissue collected (during the subjects' surgery) will also be sent to a central dermatopathologist who will be blinded to GBCA exposure and test for any possible NSF related abnormalities. These skin tissue sample(s) will be stored with the central dermatopathology laboratory.

ELIGIBILITY:
Inclusion Criteria:

SUBJECTS WHO RECEIVED MULTIHANCE or PROHANCE:

* Is scheduled to receive hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures
* Has undergone at least one MULTIHANCE or PROHANCE administration at least 1 month before his/her scheduled surgery
* Has a documented SCr for calculation of eGFR and/or documented eGFR at time of last MRI with MULTIHANCE or PROHANCE
* Provides written Informed Consent and is willing to comply with protocol requirements
* Is willing to undergo deep skin tissue sampling during scheduled hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures
* Is ≥18 years of age

SUBJECTS WITH NO EXPOSURE TO GBCA:

* Is scheduled to receive hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures
* Has no history of GBCA administration
* Provides written Informed Consent and is willing to comply with protocol requirements
* Is willing to undergo deep skin tissue sampling during scheduled hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures
* Has prior SCr and/or eGFR at time of enrollment
* Is ≥18 years of age

Exclusion Criteria:

SUBJECTS WHO RECEIVED MULTI HANCE or PROHANCE:

* Has undergone any GBCA including MULTIHANCE or PROHANCE administration less than 1 month before his/her scheduled surgery
* Has ever been suspected of, or diagnosed with, NSF
* Has been suspected or diagnosed, prior to inclusion in this study, with bone cancer or any other osteoblastic or osteoclastic disease, such as septic, infectious or ischemic disease affecting physiological bone structure that has caused the bone to be diseased, prior to inclusion in this study
* Is unable or unwilling to be examined by dermatologists or to undergo laboratory/other diagnostic evaluations should development of NSF be suspected.
* Has received any GBCA other than the one under evaluation at any time prior to inclusion in this study (e.g., a MULTIHANCE subject should not receive any other GBCA including PROHANCE)

SUBJECTS WITH NO EXPOSURE TO GBCA:

* Has received any GBCA at any time prior to inclusion in this study
* Has ever been suspected of, or diagnosed with, NSF prior to the enrollment
* Has been suspected or diagnosed with bone cancer or any other osteoblastic or osteoclastic disease, such as septic, infectious or ischemic disease affecting physiological bone structure that has caused the bone to be diseased prior to inclusion in this study
* Is unable or unwilling to be examined by dermatologists or to undergo laboratory/other diagnostic evaluations should development of NSF be suspected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled to have hip, shoulder or knee replacement surgery, limb amputations or other orthopedic surgical procedures
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Gadolinium deposition in bone and skin for non-control group | At least one month from exposure to GBCA, assessed up to a total of 36 months
  Determine the long-term gadolinium deposition in bone tissue and skin in subjects undergoing orthopedic surgery using Inductively Coupled Plasma Mass Spectroscopy (ICP-MS) in nmol gadolinium/g from surgically removed bone and skin.
Gadolinium deposition in bone and skin for control group | At any time, due to no GBCA exposure, assessed up to a total of 36 months
  Determine the long-term gadolinium deposition in bone tissue and skin in subjects undergoing orthopedic surgery using Inductively Coupled Plasma Mass Spectroscopy (ICP-MS) in nmol gadolinium/g from surgically removed bone and skin.

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No